CLINICAL TRIAL: NCT07148908
Title: The Effects of Animal- and Microbial-based Protein Sources on Whole-body Protein Metabolism in Healthy Adults
Brief Title: Animal and Microbial-based Dietary Protein Efficiency in Adults
Acronym: YPQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Moore (Other)
Collaborators: Lesaffre International (Industry)
Responsible Party: Sponsor-Investigator, Daniel Moore, Principal Investigator, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REB00048239
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Protein Metabolism
Keywords: Protein quality; protein metabolism; stable isotopes; protein oxidation; indicator amino acid oxidation; protein synthesis

STUDY DESIGN:
Intervention Model Description: Single-blind randomized, counterbalanced design
  Thirteen healthy young (18-45 years of age, at least 6 females and 6 males) will be subjected to a non-invasive 13CO2 breath-test based on the indicator amino acid oxidation method and urine collections following hourly ingestion of protein test beverages (whey, yeast, and collagen randomized by trials).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yeast Protein Supplement (Experimental): Participants will be consuming test beverage composed of yeast protein and their whole-body protein metabolism will be determined over the subsequent 8 hours.
  Interventions: Dietary Supplement: Yeast Protein Supplement
- Whey Protein Isolate Supplement (Active Comparator): Participants will be consuming test beverage composed of whey protein isolate and their whole-body protein metabolism will be determined over the subsequent 8 hours.
  Interventions: Dietary Supplement: Whey Protein Isolate Supplement
- Collagen Hydrolysate Supplement (Active Comparator): Participants will be consuming test beverage composed of collagen protein and their whole-body protein metabolism will be determined over the subsequent 8 hours.
  Interventions: Dietary Supplement: Collagen Hydrolysate Supplement

INTERVENTIONS:
Dietary Supplement: Yeast Protein Supplement — Each protein will be consumed at 0.9g/kg/d in n=8 hourly drinks
  Arms: Yeast Protein Supplement
Dietary Supplement: Whey Protein Isolate Supplement — Each protein will be consumed at 0.9g/kg/d in n=8 hourly drinks
  Arms: Whey Protein Isolate Supplement
Dietary Supplement: Collagen Hydrolysate Supplement — Each protein will be consumed at 0.9g/kg/d in n=8 hourly drinks
  Arms: Collagen Hydrolysate Supplement

SUMMARY:
Given the relatively high carbon footprint and sustainability of animal-based proteins, there is a growing interest in determining the nutritional quality non-animal-based protein sources. The overall objective of this investigation is to examine the impact of different animal and microbial-based protein sources to support whole body protein synthesis in adults. To do this, investigators will employ a 'breath test' method developed in our laboratory as well as urine sampling. The results of this study will allow us to better understand the impact of dietary protein quality for maintaining health and body protein mass in adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male and female, recreationally-active participants.
* Healthy will be defined as screened by the PAR-Q+ (Appendix B) and The Physical Activity Readiness Questionnaire (Appendix C).
* Participants will be aged 18-45 years old.
* Participants are willing to abide by the compliance rules of this study.
* Self-reported regular menstrual cycle (25-35d) within the last 3 months (female participants).
* Use of monophasic combined oral contraceptives (COC) containing 21 active pills (e.g., Yaz, Marvelon, Cyclen, etc.; the brand of COC will be recorded) (female participants).

Exclusion Criteria:

* Inability to adhere to any of the compliance rules judged by principal investigator (e.g. dairy protein or yeast allergy).
* Self-reported regular tobacco use.
* Self-reported illicit drug use (e.g., growth hormone, testosterone, etc.).
* Individuals who have participated in studies within the past year involving any of the stable isotopes in the study.
* Use of multiphasic COCs due to the difficulty of controlling for hormonal fluctuations in such formulations (female participants).
* Use of COCs containing >21 active pills per cycle due to potential differences in their effect on metabolism (female participants).
* Use of other forms of hormonal contraception (e.g., progestin-only pill, hormonal IUD, intravaginal ring) (female participants).
* Not currently or previously (in the past 6 months) on a vegan diet

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Phenylalanine excretion (umol/kg/h) | 8 hours
  Whole body phenylalanine excretion determined from the product of breath 13CO2 enrichment and carbon dioxide production rate (VCO2).
Phenylalanine oxidation (umol/kg/h) | 8 hours
  Whole-body phenylalanine oxidation determined from the correction of phenylalanine excretion by the phenylalanine precursor enrichment determined from urine enrichment over the 8 hour measurement period.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinesiology & Physical Education, Toronto, Ontario, Canada